CLINICAL TRIAL: NCT07221123
Title: A Feasibility and Acceptability Study Testing Two Types of Smell Exposure Interventions in Middle-Aged Older Adults With HIV
Brief Title: Boosting Olfactory and Sensory Training Study (BOOST)
Acronym: BOOST
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, David Vance, PhD, University Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB - 300013575; UAB (Other: UAB)
Record Dates: First submitted 2025-09-23; First posted 2025-10-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-10

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Olfactory Training

STUDY DESIGN:
Intervention Model Description: This feasibility study employs a 2-group pre-post experimental design of 80 middle-aged (40+) and older adults with cognitive complaints including: 1) a home-based Smell Training Group consisting of 8 weeks of engaging in smelling four odorants 2x/day (enroll 40, n=30 with attrition); and 2) a home-based Overnight Diffuser Group consisting of 8 weeks of engaging in using scent diffuser while one sleeps (enroll 40, n=30 with attrition)
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Smell Training Group (Experimental): We are adopting the usual smell training approach from the literature.23-32 A standard smell training kit (i.e., MOXĒ) will be used that contains the four basic odorants across the "odor prism" - i) flowery (e.g., rose), ii) resinous (e.g., eucalyptus), iii) aromatic (e.g., cloves), and iv) fruity (e.g., lemon). Participants will be instructed to sniff each of the odorant vials/bottles for 10-20 seconds twice a day (morning and evening), for the next 8 weeks. A structured daily diary will be provided for them to record observations of the experience, memories the odorants may evoke, and any side effects experienced (i.e., headache, euphoria, light headedness, phantosmia, nasal irritation).
  Interventions: Other: Standard Smell Training Group
- Overnight Diffuser Group (Experimental): This group will received a odorant diffuser and 7 essential oil odorant (rose, orange, eucalyptus, lemon, peppermint, rosemary, and lavender) from the Essential Oil Company (Portland, OR). Participants will receive instruction on how to set it up, and with a diary of keeping track of its use.
  Interventions: Other: Overnight Diffuser Grou

INTERVENTIONS:
Other: Standard Smell Training Group — We are adopting the usual smell training approach from the literature.23-32 A standard smell training kit (i.e., MOXĒ) will be used that contains the four basic odorants across the "odor prism" - i) flowery (e.g., rose), ii) resinous (e.g., eucalyptus), iii) aromatic (e.g., cloves), and iv) fruity (e.g., lemon). Participants will be instructed to sniff each of the odorant vials/bottles for 10-20 seconds twice a day (morning and evening), for the next 8 weeks. A structured daily diary will be provided for them to record observations of the experience, memories the odorants may evoke, and any side effects experienced (i.e., headache, euphoria, light headedness, phantosmia, nasal irritation).
  Other Names: olfactory training; smell training
  Arms: Standard Smell Training Group
Other: Overnight Diffuser Grou — This group will received a odorant diffuser and 7 essential oil odorant (rose, orange, eucalyptus, lemon, peppermint, rosemary, and lavender) from the Essential Oil Company (Portland, OR). Participants will receive instruction on how to set it up, and with a diary of keeping track of its use.
  Other Names: aromotherapy; smell training
  Arms: Overnight Diffuser Group

SUMMARY:
The goal of this study is to examine two types of olfactory interventions (olfactory training vs overnight odor diffuser) in adults with HIV.

The two research questions are:

1. Determine if participants find the intervention acceptable and assess feasibility of the study.
2. Determine if the intervention improves olfactory function and cognitive function.

Participants will come to our office and be administered the baseline battery of questions including olfactory and cognitive performance tests. Then they will be randomized and sent home with one of the two interventions (below) in which they will engage in it for 8 weeks, after which they come back to our office for the posttest battery of questions including olfactory and cognitive performance test.

1. Olfactory Training at Home -- 4 scents in which they will smell twice a day for 8 weeks.
2. Overnight Diffuser Group -- a single scent diffuser that participants will turn on while they sleep and use for 8 weeks.

DETAILED DESCRIPTION:
Overall A pre-post two-group experimental design will be used. Participants will be recruited from the UAB 1917 HIV/AIDS Clinic which has a patient population of +3,900 and is the largest HIV medical provider within 100 miles. Participants will be recruited via two ways: 1) flyers posted in the UAB 1917 HIV/AIDS Clinic and 2) via 1917/CINIC participant list of participants who indicated and consented they are would like to be called for recruitment to studies (a technique used before and approved in other UAB IRB studies). Eligible participants will be consented at the UAB where a ~2 hr baseline assessment will be administered. Stratified random assignment will ensure an equal number of participants in each group by gender and smoking status. Men tend to have more olfactory dysfunction than women; therefore, it is important to control for gender upfront in the methodology. After training, participants will complete a posttest assessment.

Recruitment and Retention Procedures

Flyers. Flyers advertising the study will be provide to the UAB 1917 Clinic which they can hang or post electronically on their monitors.

Electronic Medical Record Query Using CNICS EMR Data Eligibility queries may be conducted using the CFAR Network of Integrated Clinical Systems (CNICS) EMR data. Specifically, CNICS participants (which comprise over 90% of UAB 1917 Clinic patients) have consented to be contacted to gauge interest in future studies. The Research Informatics Services Center (RISC) will provide us a list of patients meeting basic criteria (e.g., based on age, last clinic data, free from major comorbidities), and we will then contact participants directly and tell them about the study and screen them over the phone as we are doing in another active study protocol (RISC - IRB-300008740). When the study concludes, we will also utilize RISC to yield a CNICS dataset for enrolled participants which will include basic health and HIV data (e.g., viral load).

Telephone Screen A brief telephone screening interview will be used to ensure that participants meet study inclusion/exclusion criteria. If participants meet entry criteria, they will be scheduled for a visit; appointment letters will indicate that if they develop a cold, flu, or other condition causing nasal obstruction in the interim, their appointment will be rescheduled. The appointment letter will instruct participants to refrain from eating highly aromatic foods (e.g., garlic) and abstain from liquor within 24 hrs of the appointment since these could affect olfactory tests. Thus, participants will review a signs and symptoms checklist to ensure they still meet study criteria. If they indicate they do not currently meet study criteria, they will be encouraged to participate when their situation changes. Once eligibility is confirmed, participants will sign an IRB approved consent form.

Inclusion Criteria. Participants (men & women) must be 40+ years and have cognitive complaints. PWH 40 years of age and older are targeted due to the greater prevalence of cognitive complaints with middle and older age.89 Because the study instruments are standardized in English, participants must be proficient in English.

Exclusion Criteria. Because the following conditions can affect chemosensory (smell & taste) abilities, participants will be excluded if they have any of the following: a sinus infection (within the past 3 months), thrush, candidiasis, pregnant, current cold or flu, hay fever, asthma, nasal allergies, opportunistic infections (including COVID-19) within the past 3 months, or current nasal obstruction condition. Participation requires ~8 weeks and in-person visits, participants living beyond 60 miles away from the center will be excluded. Participants living in unstable housing (e.g., shelter) or with significant neuro-comorbidities (e.g., schizophrenia) will be excluded. Other conditions (e.g., legally blind/deaf, currently undergoing radiation or chemotherapy, or a history of significant brain trauma) that could impact olfactory and cognitive testing also necessitate exclusion. These criteria are typical of neuroHIV and olfaction studies.

Rationale for Including Smokers. Furthering the ecological validity, we will include tobacco smokers to make the study more generalizable. Our olfactory study revealed that it was difficult to recruit non-smokers given that the high prevalence of smoking in PWH (39% current and 29% former smokers).95 In our past R01 study of 260 PWH 40+, 53% were current smokers. Contrary to expectations, smoking is not associated with changes in olfaction. In fact, in our prior study, cigarettes smoked per day was not related to any cognitive or olfactory measures. In this case, smoking appears not to confound the study results. Confirming this, studies affirm that habitual smokers do not experience olfactory declines as commonly thought and actually smoking may preserve olfaction.

Recruitment and Retention Strategy. As has been effective in our prior studies, flyers will be used to recruit patients from our HIV/AIDS Clinic. Other recruitment/retention strategies include: 1. Compensation will be provided ($50 at baseline & $50 for posttest assessment, $20 to return the completed smell training/smell exposure dairy; and $5 for each weekly questionnaire completed). 2. Telephone calls will be made and reminder letters will be sent before the scheduled visit. 3. Secondary contact information will be collected to follow up with lost participants.

Intervention Protocol At the end of the baseline visit, we will randomize the participants. The research assistant will provide the participant with the smell exposure materials, diary, and instructions.

Standard Smell Training Group - We are adopting the usual smell training approach from the literature. A standard smell training kit (i.e., MOXĒ) will be used that contains the four basic odorants across the "odor prism" - i) flowery (e.g., rose), ii) resinous (e.g., eucalyptus), iii) aromatic (e.g., cloves), and iv) fruity (e.g., lemon). Participants will be instructed to sniff each of the odorant vials/bottles for 10-20 seconds twice a day (morning and evening), for the next 8 weeks. A structured daily diary will be provided for them to record observations of the experience, memories the odorants may evoke, and any side effects experienced (i.e., headache, euphoria, light headedness, phantosmia, nasal irritation).

Overnight Diffuser Group40 - This group will received a odorant diffuser and 7 essential oil odorant (rose, orange, eucalyptus, lemon, peppermint, rosemary, and lavender) from the Essential Oil Company (Portland, OR). Participants will receive instruction on how to set it up, and with a diary of keeping track of its use.

Instruments (Baseline and Posttest) Because participants will be recruited through the UAB 1917 (HIV/AIDS) Clinic, the following information will be available for analysis from the electronic medical records through the CFAR Statistical Core; body mass index, most recent t-cell count, viral load, cholesterol, and serum albumin levels that correspond most closely to their study visit. Testing will be reviewed and observed every quarter to prevent drift in the protocol.

Demographic, Background, and Covariate Measures (*Baseline Only)

* Demographic Questionnaire - Used to gather basic background characteristics (e.g., gender, ethnicity, etc). ( 2 min.)
* Wide Range Achievement Test-3 (WRAT-3) - Used to determine educational quality. (2 min.) Centers for Epidemiological Studies - Depression (CES-D) scale measures how often (participants acknowledge 20 verbal depressive symptoms. Cronbach's α is very good at 0.88. (2 min.) Cognitive Complaints - Cognitive Failures Questionnaire (CFQ) - CFQ assesses common everyday cognitive complaints one may have such as in memory (e.g., "Do you forget where you put something?"). (3 min.) Health-Related Quality of Life - Medical Outcomes Study - HIV - Short Form (SF-35) - The SF-35 includes one multi-item scale that assesses 8 health-related quality of life concepts. Cronbach's alphas for the concepts are excellent (<0.85). (10 min.)
* HIV History/Status - Used to assess current HIV status (i.e., viral load) and general HIV infection history. (2 min.) Addiction Severity Index (ASI) - A widely used, gold standard measure of alcohol and drug use. (4 min.)
* HIV History/Status - Used to assess current HIV status (i.e., viral load) and general HIV infection history. (2 min.)

Feasibility and Acceptability Measures A training diary will be given to participants to help them keep track of their engagement in the protocol. It will have simple check boxes for ease of use as well as space to write comments/observations. Participants will also receive a weekly call from the Principal Investigator/Research Assistant and be asked to recall how many days in the past seven have they engaged in the intervention as directed; field notes will be taken to document protocol processes that aid or interfere with the study. In addition, daily text messages Monday-Friday will be sent as reminders to encourage use of the Smell Training/Smell Exposure protocol. At the Posttest Visit after use of the Smell Exposure protocols, participants will also be asked a series of questions about what they liked and did not like about using the smelling training protocols. Many of these questions are open-ended and will be coded and used in qualitative analyses. This information will be used to determine the barriers and facilitators of the intervention. Treatment adherence will be measured by daily diaries, and posttest assessment. Study attrition will also be monitored. Many of these protocols have been used in our prior studies to document treatment fidelity and feasibility.

Olfactory Training Satisfaction Questionnaire (posttest only) - Used to assess likes/dislikes of the intervention); both quantitative questions and qualitative (i.e., open-ended responses) data are gathered as has been used in our previous cognitive intervention studies to evaluate feasibility and acceptability. (10 min.)

Side Effect Questionnaire (posttest only) - We will provide a list of potential good and bad side effects of engaging in smell training/smell exposure. Participants will indicate which ones they experienced, how often, and to what degree it affected them. (5 min.) Daily Diaries (treatment monitoring) - This data collection method may provide insights into some of the experiences of those engaged in the smell training/smell exposure. It is also a source of convergent validity concerning adherence.

Attrition & Adherence Rates (after study data collection) - We will calculate the attrition rate and adherence rate of the protocol, similar to our other studies.

Olfactory (Chemosensory) Measures Smell is 10,000 times more powerful than taste, with taste being approximately 75% smell. In fact, it is the neural integration of smell and taste that produces the sensation of flavor. For these reasons, only tests of smell are used.

Smell Identification -- University of Pennsylvania Smell Identification Test (UPSIT) - The UPSIT is to smell as an eye chart is to vision and has been used extensively in the literature.115,116 Age and gender-based norms from 4,000 men and women over the lifespan have provided a percentile rank of how each participant, based on his/her sex and age, performs along a normal distribution. The UPSIT is composed of 40 test items containing 40 microencapsulated "scratch and sniff" odors. This test-retest for UPSIT is very reliable (r = 0.94). (10 min.)

Taste & Smell Questionnaire Taste and Smell Questionnaire - Heald et al. (1998) used a smell and taste questionnaire for adults with HIV. The taste section consists of nine questions that address changes in the way food tastes. The smell section consists of five questions that address changes in the sense of smell. This measure was found to be related to the SF-36 (below)108 mental health and physical health summaries (p<.01). (50 min.)

Cognitive Measures. Both mean-level cognitive functioning (e.g., domain specific and global cognitive functioning) and cognitive intra-individual variability calculations will be used to examine cognitive change.

BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning), supported by NIMH R42099964 and Digital Artefacts/UCSD) is a HIPAA compliant tablet-based cognitive assessment platform. This self-administered tool is not literacy dependent (i.e., automated audio and video instructions) and uses validated cognitive tests that are sensitive to mild-to-moderate cognitive deficits and have demonstrated good validity relative to a comprehensive standard neuropsychological test battery and test-retest reliability. The BRACE+ measures to be administered in each of the cognitive domains (i.e., executive function, etc.).

IIV Dispersion - Dispersion (IIVD) is one type of IIV that refers to variability in performance across multiple measures, such as across tests in the neuropsychological test battery (above). There are two accepted formulas: 1) the intra-individual standard deviation (iSD), and 2) the coefficient of variation (CoV) (Vance et al., submitted). Both will be calculated at baseline and posttest as an outcome variable; it is hypothesized that IIV Dispersion will decrease in those in the training groups.

IIV Inconsistency using the Connors' Continuous Performance Test - Inconsistency (IIVC) is another type of IIV that refers to variability related to a single person's performance on a single task (i.e., within task) across multiple instances or trials, such as the variability observed across a person's distribution of reaction times (RT) on a cognitive task. There are two accepted formulas: 1) the intra-individual standard deviation (iSD), and 2) the coefficient of variation (CoV) (Vance et al., submitted). These also will be calculated at baseline and posttest as an outcome variable as a measure of overall improved cognitive function. The Connor's Continuous Performance Test, Second Edition (CPT-II) is a widely accepted test of sustained/selective attention and impulsivity (10 min); it is also used to calculate IIVc.

Data Analysis Data Management and Tracking. The research assistant/study coordinator will double-key enter de-identified questionnaire responses into an encrypted, password protected (front and back end) electronic database called REDCap (Research Electronic Data CAPture). The PI will follow-up and resolve any data queries resulting from the quality control process.

Analysis Plan. Data will be analyzed using SPSS, R, and/or SAS for simple pre-post analyses (i.e., ANCOVA). From this, effect sizes can be calculated that can be used in power analyses for future grant submissions. Also, the qualitative data will be used to modify the intervention and improve on tracking and adherence to the protocol for future studies.

ELIGIBILITY:
Inclusion Criteria:

* Participants (men & women) must be 40+ years
* have cognitive complaints.
* must be proficient in English

Exclusion Criteria:

* a sinus infection (within the past 3 months), thrush, candidiasis, pregnant, current cold or flu, hay fever, asthma, nasal allergies, opportunistic infections (including COVID-19) within the past 3 months, or current nasal obstruction condition.
* Participation requires ~8 weeks and in-person visits, participants living beyond 60 miles away from the center will be excluded.
* Participants living in unstable housing (e.g., shelter) or with significant neuro-comorbidities (e.g., schizophrenia) will be excluded.
* Other conditions (e.g., legally blind/deaf, currently undergoing radiation or chemotherapy, or a history of significant brain trauma) that could impact olfactory and cognitive testing also necessitate exclusion.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
FEASIBILITY & ACCEPTABILITY | From enrollment to the end of treatment at 8 weeks
  A training diary will be given to participants to help them keep track of their engagement in the protocol. It will have simple check boxes for ease of use as well as space to write comments/observations. Participants will also receive a weekly call from the Principal Investigator/Research Assistant and be asked to recall how many days in the past seven have they engaged in the intervention as directed; field notes will be taken to document protocol processes that aid or interfere with the study. In addition, daily text messages Monday-Friday will be sent as reminders to encourage use of the Smell Training/Smell Exposure protocol. At the Posttest Visit after use of the Smell Exposure protocols, participants will also be asked a series of questions about what they liked and did not like about using the smelling training protocols. Many of these questions are open-ended and will be coded and used in qualitative analyses.

SECONDARY OUTCOMES:
OLFACTION | From enrollment to the end of treatment at 8 weeks
  University of Pennsylvania Smell Identification Test (UPSIT) - The UPSIT is to smell as an eye chart is to vision and has been used extensively in the literature.115,116 Age and gender-based norms from 4,000 men and women over the lifespan have provided a percentile rank of how each participant, based on his/her sex and age, performs along a normal distribution. The UPSIT is composed of 40 test items containing 40 microencapsulated "scratch and sniff" odors. This test-retest for UPSIT is very reliable (r = 0.94). (10 min.)
  Taste and Smell Questionnaire - Heald et al. (1998) used a smell and taste questionnaire for adults with HIV. The taste section consists of nine questions that address changes in the way food tastes. The smell section consists of five questions that address changes in the sense of smell. This measure was found to be related to the SF-36 (below) mental health and physical health summaries (p<.01). (50 min.)
COGNITION | From enrollment to the end of treatment at 8 weeks
  BRACE+ (BrainBaseline Assessment of Cognition and Everyday Functioning), supported by NIMH R42099964 and Digital Artefacts/UCSD) is a HIPAA compliant tablet-based cognitive assessment platform. This self-administered tool is not literacy dependent (i.e., automated audio and video instructions) and uses validated cognitive tests that are sensitive to mild-to-moderate cognitive deficits and have demonstrated good validity relative to a comprehensive standard neuropsychological test battery and test-retest reliability. The BRACE+ measures to be administered in each of the cognitive domains (i.e., executive function).
  IIV Inconsistency using the Connors' Continuous Performance Test - Inconsistency (IIVC) is another type of IIV that refers to variability related to a single person's performance on a single task (i.e., within task) across multiple instances or trials, such as the variability observed across a person's distribution of reaction times (RT) on a cognitive task.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This is a small internal pilot grant used to generate data for grant submission and for secondary data use for a PHD student at the same institution.

REFERENCES:
- [Result] Kamath V, Del Bene VA, Collette C, Jacob A, Fazeli PL, Vance DE. A Pilot Study of Self-Rated and Psychophysical Olfactory Dysfunction in Men Living with HIV. Chemosens Percept. 2022;15(2):175-184. doi: 10.1007/s12078-022-09305-x. Epub 2022 Nov 10. PMID 36406043
- [Result] Vance D, Burrage J. Chemosensory declines in older adults with HIV: identifying interventions. J Gerontol Nurs. 2006 Jul;32(7):42-8. doi: 10.3928/00989134-20060701-06. PMID 16863045
- [Result] Vance DE, Del Bene VA, Kamath V, Frank JS, Billings R, Cho DY, Byun JY, Jacob A, Anderson JN, Visscher K, Triebel K, Martin KM, Li W, Puga F, Fazeli PL. Does Olfactory Training Improve Brain Function and Cognition? A Systematic Review. Neuropsychol Rev. 2024 Mar;34(1):155-191. doi: 10.1007/s11065-022-09573-0. Epub 2023 Feb 2. PMID 36725781
- [Result] Vance DE, Cody SL, Nicholson WC, Cheatwood J, Morrison S, Fazeli PL. The Association Between Olfactory Function and Cognition in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2019 Sep-Oct;30(5):e144-e155. doi: 10.1097/JNC.0000000000000086. PMID 31259847
- [Result] Vance DE, Cody SL, Nicholson C, Cheatwood J, Morrison S, Fazeli PL. Olfactory Dysfunction in Aging African American and Caucasian Men With HIV: A Pilot Study. J Assoc Nurses AIDS Care. 2022 May-Jun 01;33(3):e19-e30. doi: 10.1097/JNC.0000000000000061. PMID 30676359